CLINICAL TRIAL: NCT05746026
Title: Effectiveness of Psycho-educational Program on Climate Change Distress and Risk Perception Among Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1522023
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Psycho-educational Programو Climate Change Distressو Risk Perception, Older Adults

STUDY DESIGN:
Intervention Model Description: * Session 1: introduction and basic information about Climate Change: the researcher was describing the significance of the intended educational program sessions as well as the expected aims to be met.
  * Session 3: explain climate change risks, describe and explain the impact of climate change on elder health and well-being. These consequences obviously include biological impacts and hazards to physical health and to human, also direct and indirect psychological and interpersonal impacts of climate change.
  * Session 4: teaching proper behaviors that contribute the most to climate-driving emissions.
  * Session 5: learning how adapting and coping with climate change. Adaptation includes a range of coping actions that individuals may take, as well as psychological processes
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): • The study subjects who fulfilled the inclusion criteria were interviewed individually in the garden of the clubs in order to collect the necessary data (tool I, II, III, and IV). Then, the researcher interviewed the clients in group composed of 8 older adults to implement the Psycho-educational Program . Each session taken about 30-45 minutes.
  Interventions: Behavioral: Psycho-educational Program
- Control group (Active Comparator): Control group exposed to the usual routine care
  Interventions: Behavioral: Psycho-educational Program

INTERVENTIONS:
Behavioral: Psycho-educational Program — This program consisted of five (5) sessions during two weeks.
  * Session 1: introduction and basic information about Climate Change
  * Session 2: causes and factors that contribute to climate change by humans and nature
  * Session 3: explain climate change risks, describe and explain the impact of climate change on elder health and well-being.
  * Session 4: teaching proper behaviors that contribute the most to climate-driving emissions.
  * Session 5: learning how adapting and coping with climate change. Adaptation includes a range of coping actions that individuals may take, as well as psychological processes (e.g. emotion management, problem solving, and cognitive reframing responses) that influence reactions to (and preparations for) adverse impacts of climate change, including chronic environmental conditions and extreme events.

SUMMARY:
Research design The study followed a quasi-experimental study with two groups (study and control group) with a pre-test and post-test.

Setting:

This study was conducted at three elderly clubs at Damanhour city, El-Behaira Governorate, Egypt. These clubs are affiliated to the Ministry of Social Solidarity, Egypt namely Ahbab Allah, Alfady, and Alrabie Clubs. These clubs opens seven days per week from 9 am to 12 pm. The total attendance rate of older adults in these clubs amounted to 213; 93 older adults in Alfady Club, 70 in Ahbab Allah Club and 50 older adults in Alrabie Club.

DETAILED DESCRIPTION:
* An Official letter from the Faculty of Nursing, Damanhour University was directed to the director of the Ministry of Social Solidarity in El -Behira governorate to obtain permission to conduct the study, then to the directors of the three elderly clubs in Damanhour city to obtain their approval to carry out the study.
* A Socio-Demographic Data and clinical Structured Interview Schedule (tool II) was developed by the researchers based on review of related literature. The Arabic version of tool I (Mini-Mental State Examination) and tool IV (Risk Perception Scale) were used in this study.
* The study subjects who fulfilled the inclusion criteria were interviewed individually in the garden of the clubs in order to collect the necessary data (tool I, II, III, and IV). Then, the researcher interviewed the clients in group composed of 8 older adults to implement program. Each session taken about 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years and above.
2. Able to communicate effectively.
3. Did not have malignancies or psychiatric diseases.

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Climate Change Distress and Impairment Scale (CC-DIS): | 2 weeks
  It was developed by Hepp et al., (2022) to assesses level of different types of affect in response to climate (Anger, Anxiety, and Sadness) in addition, climate change impairment (CCI) that cover general, social, and work related impairment. It consists of 23 items with 9 statements (3, 5, 7, 10, 13, 15, 17, 20, and 21) from the scale are negatively stated and reversely scored. Factor analysis of the scale yielded four factors. Factor I consist of 5 statements (1, 4, 7, 10, and 13) describing anger. Factor II consisting of 5 statements (2, 5, 8, 11, and 15) that measure anxiety. Factor III, consisting of 5 statements (3, 6, 9, 12, and 14) is related to sadness, and finally 8 statements measure impairment.
Risk Perception Scale: | 2 weeks
  The scale was adapted from van der Linden (2015) who based his measurements on previous work by Bord et al. (2000) and Leiserowitz (2006). It was translated into Arabic language by Elshirbiny (2018) and proved to be valid.
  The scale comprises 8 statements. In the first question respondents were asked to rate how likely they thought it was that they would personally experience serious threats to their wellbeing. The second question asked how likely it was that climate change would have harmful long-term impacts on society. The two questions used a 7-point scale ranging from very unlikely (1) to very likely (7). The following four questions asked the respondents to rate how serious a threat climate change was to the natural environment, how serious the current impacts of climate change around the world were, and how serious the threat of climate change was to them personally and to Egypt. A 7-point scale was used ranging from not serious at all (1) to very serious (7).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: No